CLINICAL TRIAL: NCT06562062
Title: Radiological Outcomes of Modified Extra-articular Lateral Column Lengthening Procedure for Correction of Adult Acquired Flexible Flatfoot Deformity
Brief Title: Radiological Outcomes of Modified Extra-articular LCL
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hosam Eldeen Kamal Mohamed, Hosam Eldeen Kamal Mohamed, Assiut University
Other Study IDs: Extra-articular LCL of AAFFD
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Adult Acquired Flexible Flatfoot Deformity After Failure of Conservative Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extra-articular Lateral Column Lengthening Procedure — Lateral column lengthening (LCL), originally described by Evans, is an established procedure to correct stage II adult acquired flatfoot deformity (AAFD). However, the relative position between the facets is violated, and other problems may include nonunion, malunion, and calcaneocuboid (CC) joint subluxation. Herein, we report a modified extra-articular technique of LCL with hockey-stick osteotomy, which preserves the subtalar joint as a whole, increases bony apposition to enhance healing ability, and preserves the insertion of the calcaneofibular ligament to stabilize the posterior fragment to promote adduction of the forefoot

SUMMARY:
To assess radiological and functional outcomes of modified extra-articular lateral column lengthening procedure for correction of adult acquired flexible flatfoot deformity

DETAILED DESCRIPTION:
Measurement of

1. Calcencal pitch : This angle is formed on a weight-bearing lateral foot radiograph between the calcaneal Inclination axis and the supporting horizontal surface(10), normal ranges of between 10-25° and 20-30 have Been proposed(11)
2. Meary's angle: It is the angle between a line drawn along the longitudinal axis of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) , typically', Meary's angle is 0°, with abnormal values considered angle >4° convex upward: pes cavus , angle <-4 convex downward: pes planus, It can be used to classify the severity of deformity
3. lateral talocalceneal angle : the angle between the calcaneal inclination axis and the mid-talar axis , The lateral talocalcaneal angle should normally measure between 25 and 40°, >40° diagnoses flatfoot deformity(12)
4. Talonavicular coverage angle: it is the medial angle between ( talar head articular surface and Proximal navicular articular surface) ,Interpreting the talonavicular coverage angle (13)Normal: <7,Adult Acquired flatfoot disease: >7°

ELIGIBILITY:
Inclusion Criteria:

- 1) Age : adult ( age above 16 years old and below 65 years old

2) symptomatic flexible flat foot after failure of Conservative treatment

Exclusion Criteria:

* 1- Age: (<16,>65) years old 2 -Previous foot surgery 3- autoimmune disease
* 4 Uncontrolled blood sugar 5- Osteoprotic patient 6- Infection

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult flexible acquired flatfoot deformity which doesn't include genetic or spasmodic flatfoot deformity in children
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-08-16 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Radiological outcome & by standard erect plain x ray after 3 months | 3 months after the surgery
  Measurement of
  1. Calcencal pitch : this angle is formed on a weight-bearing lateral foot radiograph between the calcaneal Inclination axis and the supporting horizontal surface , correction angle needed ≈ 15-25°.
  2. Meary's angle: It is the angle between a line drawn along the longitudinal axis of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) , correction angle needed ≈ 0-1°.
  3. lateral talocalceneal angle : the angle between the calcaneal inclination axis and the mid-talar axis correction angle ≈ 25 and 40° .
  4. Talonavicular coverage angle: it is the medial angle between ( talar head articular surface and Proximal navicular articular surface

SECONDARY OUTCOMES:
clinical outcome by American orthopedic foot and ankle score (hindfoot | 6 months after the surgery when the patient restore his life activities maximally

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine assiut university, Asyut, Assiuu, Egypt